CLINICAL TRIAL: NCT07015073
Title: Comparative Efficacy and Tolerability of Pulsed Dye Laser and Potassium-titanyl-phosphate Laser Treatment for Capillary Malformations: Sequential Versus Single Application
Brief Title: Comparative of Sequential Application of Pulsed Dye Laser and Potassium-titanyl-phosphate Laser Treatment for Capillary Malformations Versus Single Application
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Jorge Naharro-Rodriguez, M.D., Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 232/24
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Port-Wine Stains (Capillary Malformations)
Keywords: port-wine stains; capillar malformation; laser; pulsed dye laser; KTP laser
MeSH Terms: conditions — Port-Wine Stain; Capillary Malformations, Congenital, 1 | interventions — Lasers, Dye; Lasers

STUDY DESIGN:
Intervention Model Description: Crossover Assignment (within-subject comparison of three treatment modalities on different lesion areas)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Pulsed Dye Laser (PDL) (Active Comparator): Participants will receive pulsed dye laser treatment (595 nm) on one defined area of their port-wine stain. The treatment will be administered using the VBeam Prima® system (Candela Medical) with standard clinical parameters: 10 mm spot size, 7-9 J/cm² fluence, and 0.5-3 ms pulse duration. Cryogen spray cooling will be used, and no anesthesia will be applied.
  Interventions: Device: Pulsed dye laser (PDL)
- Potassium Titanyl Phosphate Laser (KTP) (Active Comparator): Participants will receive potassium titanyl phosphate laser treatment (532 nm) on another defined area of the same lesion. Treatment will be performed using the DermaV® system (Lutronic Medical Systems) with standard parameters: 10 mm spot size, 8-11 J/cm² fluence, and 10 ms pulse duration. Cryogen spray cooling will be used; no anesthesia will be applied.
  Interventions: Device: Potassium titanyl phosphate (KTP) laser
- Sequential KTP + PDL (Experimental): Participants will receive sequential treatment on a third, anatomically matched area of their port-wine stain. The area will first be treated with the KTP laser (532 nm; DermaV® system), followed immediately by pulsed dye laser (595 nm; VBeam Prima®). Parameters for each device will match those used in the monotherapy arms. Cryogen spray cooling will be applied before each pass, without anesthesia.
  Interventions: Device: Sequential KTP + PDL laser treatment

INTERVENTIONS:
Device: Pulsed dye laser (PDL) — Treatment with a pulsed dye laser (PDL) at 595 nm using the VBeam Prima® system (Candela Medical). Parameters: 10 mm spot size, 7-9 J/cm² fluence, 0.5-3 ms pulse duration. Cryogen spray cooling is applied. No anesthesia is used. This intervention will be applied to one of the three defined regions of each participant's port-wine stain.
  Arms: Pulsed Dye Laser (PDL)
Device: Potassium titanyl phosphate (KTP) laser — Treatment with a KTP laser at 532 nm using the DermaV® system (Lutronic Medical Systems). Parameters: 10 mm spot size, 8-11 J/cm² fluence, 10 ms pulse duration. Cryogen spray cooling is applied. No anesthesia is used. This intervention will be applied to a second anatomically comparable region of the port-wine stain.
  Arms: Potassium Titanyl Phosphate Laser (KTP)
Device: Sequential KTP + PDL laser treatment — Sequential treatment of the same region with two lasers: first with KTP (532 nm, DermaV® system), then with PDL (595 nm, VBeam Prima® system). Each laser will be applied using its standard parameters: KTP (10 mm spot, 8-11 J/cm², 10 ms), followed by PDL (10 mm spot, 7-9 J/cm², 0.5-3 ms). Cryogen spray cooling is used before each pass. No anesthesia is applied. This treatment is administered to a third region of the port-wine stain.
  Arms: Sequential KTP + PDL

SUMMARY:
This prospective, non-randomized study aims to evaluate the efficacy and tolerability of treating port-wine stains (capillary malformations) using pulsed dye laser (PDL), potassium titanyl phosphate (KTP) laser, or a sequential combination of both. Each participant will receive all three treatments on different areas of the lesion. The primary outcome is improvement measured using the Investigator Global Assessment (IGA) scale. Secondary outcomes include pain (VAS), local adverse events, and patient satisfaction.

DETAILED DESCRIPTION:
Port-wine stains (PWS), also known as capillary malformations, are congenital vascular anomalies affecting approximately 0.3-0.5% of newborns. These lesions, often located on the face and neck, tend to darken and thicken over time, potentially leading to psychosocial distress and reduced quality of life. Pulsed dye laser (PDL) therapy has long been the standard of care, utilizing selective photothermolysis to target dilated capillaries. Despite its safety and effectiveness, complete clearance is achieved in only 10-20% of cases.

Recently, long-pulsed potassium titanyl phosphate (KTP) lasers operating at 532 nm have emerged as viable options for vascular lesions, offering greater spot sizes, variable pulse durations, and integrated cryogen cooling systems that allow deeper and more consistent energy delivery. Clinical experience suggests that combining PDL and KTP treatments sequentially may enhance treatment outcomes, especially in resistant PWS, yet no controlled study has directly compared this approach to either treatment in isolation.

This prospective, single-center, non-randomized clinical trial aims to compare the efficacy, safety, and patient satisfaction of PDL (595 nm), KTP (532 nm), and sequential KTP followed by PDL in adults with PWS. Each lesion will be divided into three anatomically comparable areas, each receiving a different treatment modality. All treatments will be administered with cryogen spray cooling and without anesthesia, according to current clinical practice.

The primary endpoint is improvement at 6 weeks based on the Investigator Global Assessment (IGA) scale, evaluated by three blinded dermatologists. Secondary outcomes include pain during treatment (VAS), adverse events at 48 hours, and patient satisfaction scores. A total of 30 patients will be enrolled to ensure adequate statistical power and account for potential dropouts.

This study seeks to provide evidence supporting the optimal laser treatment strategy for PWS, potentially improving clinical outcomes and guiding future protocols.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Fitzpatrick skin types I-IV
* Presence of port-wine stain

Exclusion Criteria:

* Open wounds in treatment area
* Pregnancy
* Nearby metal implants
* Photodermatoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in lesion appearance measured by Investigator Global Assessment (IGA) | 6 weeks after treatment
  The IGA is a 5-point scale ranging from 0 (no changes) to 4 (complete or near-complete clearance). It will be assessed by three blinded dermatologists comparing standardized clinical photographs of each treated area. The outcome will be reported as the mean IGA score per treatment modality.

SECONDARY OUTCOMES:
Pain score during laser treatment (VAS) | Immediately after the procedure
  Participants will rate their pain during each treatment using a Visual Analog Scale (VAS) from 0 (no pain) to 10 (maximum imaginable pain).
Local events at 48 hours | 48 hours after treatment
  Presence of local side effects such as edema, purpura, and crusting will be documented clinically by the investigators.
Patient satisfaction score | 6 weeks after treatment
  Patients will rate their satisfaction with each treated area on a scale from 0 (not satisfied at all) to 6 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Ramon y Cajal University Hospital, Madrid, Spain, Spain

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data (IPD). The collected data will be coded and stored securely, accessible only to the investigators and regulatory authorities, in compliance with the General Data Protection Regulation (GDPR) and Spanish data protection law. Any future data sharing will be limited to aggregated, de-identified results published in scientific journals or presented at conferences, with no identifiable personal information disclosed.